CLINICAL TRIAL: NCT01254318
Title: Temporal Realistic Assessment of the Fungal Infection Incidence Across Canada for High Risk Subjects With Hematological Disease (TRAFIC)
Brief Title: Assessment of the Fungal Infection Incidence Across Canada for High Risk Participants With Hematological Disease (P07501)
Acronym: TRAFIC
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: P07501; MK-5592-071 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-11-05; First posted 2010-12-06 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Mycoses; Leukemia
Keywords: hematological malignancy; fungal infection; leukemia
MeSH Terms: conditions — Mycoses; Leukemia; Hematologic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants at high risk for IFI: Participants will be considered high risk if they are undergoing high dose chemotherapy for leukemia. This includes, but is not limited to participants with acute myelogenous leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome. Participants are also considered to be at high risk for IFI if they have undergone allogeneic hematopoietic stem-cell transplantation.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — Health-care interventions will be recorded; no additional procedures outside the standard of care will be required.

SUMMARY:
This will be a retrospective study that includes retrospective chart reviews at major institutions across Canada. The intent of the study is to generate both regional and national incidence data for non-Candida invasive fungal infections (IFI) in high risk participants. The study will include participants receiving stem cell transplant and high dose chemotherapy treatment for leukemia.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for study inclusion, the participant must have:
* A hematological malignancy requiring high dose chemotherapy with or without bone marrow transplant

Exclusion Criteria:

* The participant is not eligible for study inclusion if:
* Their IFI is not related to hematological malignancies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants at high risk for IFI at medical institutions in Canada
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hematologic malignancy requiring high dose chemotherapy with or without stem cell transplant were selected from a single tertiary care center in Canada.
Groups:
- Participants at High Risk for IFI: Participants were considered high risk for IFI if they were undergoing high dose chemotherapy for leukemia. This includes, but is not limited to participants with acute myelogenous leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome. Participants were also considered to be at high risk for IFI if they had undergone allogeneic hematopoietic stem cell transplantation.
Period: Overall Study
Arm/Group | Participants at High Risk for IFI
Started | 130 (Alive at start of study)
Completed | 78 (Alive at end of study)
Not Completed | 52
Not completed — Lost to Follow-up | 5
Not completed — Death | 47

BASELINE CHARACTERISTICS:
Groups:
- Participants at High Risk for IFI: Participants were considered high risk for IFI if they were undergoing high dose chemotherapy for leukemia. This includes, but is not limited to participants with acute myelogenous leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome. Participants were also considered to be at high risk for IFI if they had undergone allogeneic hematopoietic stem-cell transplantation.
Arm/Group | Participants at High Risk for IFI
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.28 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-Candida Invasive Fungal Infections at a Single Institution
Description: Data were extracted from participant hospital records from the time of initiating chemotherapy or conditioning regimen for their stem cell transplant (index date) until one year post-index date, in order to determine the percentage of high risk participants with non-Candida invasive fungal infections.
Time Frame: 365 days
Population: All enrolled participants who received stem-cell transplant and high dose chemotherapy for leukemia.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants at High Risk for IFI
Number analyzed (Participants) | 130
Percentage of participants | 32.3 [24.4 to 41.1]

2. Secondary Outcome: Percentage of Participants With a Specific Fungal Pathogen at a Single Institution
Description: Data were extracted from participant hospital records from the time of initiating chemotherapy or conditioning regimen for their stem cell transplant (index date) until one year post-index date, in order to determine the percentage of participants with a specific fungal pathogen.
Time Frame: 365 days
Population: All enrolled participants who received stem cell transplant and high dose chemotherapy for leukemia.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants at High Risk for IFI
Number analyzed (Participants) | 130
Percentage of participants
  Aspergillus | 8.5
  Fusarium | 1.5
  Penicillium | 0.8
  Missing | 21.5

3. Secondary Outcome: Percentage of Participants With Invasive Fungal Infections in Canada
Description: Data were to be extracted from participant hospital records from 5-9 centers across Canada starting from the time of initiating chemotherapy or conditioning regimen for their stem cell transplant (index date) until one year post-index date, in order to determine the percentage of high risk participants with non-Candida invasive fungal infections.
Time Frame: 365 days
Population: Whereas enrollment at 5-9 centers in Canada was planned, this was not accomplished, as data were only collected from a single institution in Canada.
Arm/Group | Participants at High Risk for IFI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events were not collected during this study.
Arm/Group | Participants at High Risk for IFI
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator and Institution agree to provide 45 days written notice to Sponsor prior to submission for publication or presentation to permit Sponsor to review drafts of abstracts and manuscripts for publication which report any results arising out of the Study.